CLINICAL TRIAL: NCT05732805
Title: A Double-Blind Placebo-Controlled Comparative Randomized Clinical Study of the Efficacy and Safety of BCD-217 (Nurulimab + Prolgolimab) Followed by Anti-PD-1 Compared to Anti-PD-1 Monotherapy as First-Line Treatment in Subjects With Unresectable/Metastatic Melanoma
Brief Title: A Clinical Study of BCD-217 (Nurulimab + Prolgolimab) Followed by Anti-PD-1 Compared to Anti-PD-1 Monotherapy as First-Line Treatment in Subjects With Unresectable/Metastatic Melanoma
Acronym: OCTAVA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-217-2
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Melanoma; Melanoma (Skin); Melanoma Stage III; Melanoma Stage IV; Melanoma Unresectable; Melanoma Metastatic; Melanoma Advanced
Keywords: PD-1; CTLA-4; prolgolimab; nurulimab; immunotherapy; checkpoint inhibitors; CPI; programm death; cytotoxic T-lymphocyte-associated protein
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-217 (nurulimab + prolgolimab) (Experimental): BCD-217 followed by prolgolimab 1 mg/kg monotherapy.
  Interventions: Biological: BCD-217; Biological: BCD-100; Biological: Placebo
- BCD-100 (prolgolimab) (Active Comparator): Prolgolimab monotherapy.
  Interventions: Biological: BCD-100; Biological: Placebo

INTERVENTIONS:
Biological: BCD-217 — Subject recieves BCD-217 0.2 mL/kg, which is equivalent to 1 mg/kg nurulimab + 3 mg/kg prolgolimab, as an intravenous infusion once every 3 weeks (Q3W) simultaneously with placebo, a total of 4 intravenous infusions. Beginning with the 5th infusion, subjects are switched to prolgolimab 1 mg/kg monotherapy once every 2 weeks (Q2W).
  Other Names: nurulimab+prolgolimab
  Arms: BCD-217 (nurulimab + prolgolimab)
Biological: BCD-100 — Subject recieves prolgolimab 3 mg/kg as an intravenous infusion once every 3 weeks (Q3W) simultaneously with placebo, a total of 4 intravenous infusions. Beginning with the 5th infusion, subjects are switched to prolgolimab 1 mg/kg monotherapy once every 2 weeks (Q2W).
  Other Names: prolgolimab; Forteca
Biological: Placebo — Placebo

SUMMARY:
The aim of study is to investigate the efficacy, safety, immunogenicity, pharmacokinetics, and pharmacodynamics of BCD-217 followed by prolgolimab monotherapy versus prolgolimab monotherapy as first-line therapy in subjects with unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
This study is designed as a phase III, randomized, double-blind, placebo-controlled study.

After the stratification procedure, subjects are randomized in a 1:1 ratio into 2 groups:

* BCD-217 + placebo (4 doses) → prolgolimab (BCD-217 group)
* Prolgolimab + placebo (4 doses) → prolgolimab (BCD-100 monotherapy group)

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and the subject's ability to comply with the requirements of the clinical study protocol;
2. Age ≥18 years at the time of signing the informed consent form;
3. Histologically confirmed melanoma (with available documented evidence of relevant investigations);
4. Untreated unresectable stage III melanoma or untreated metastatic (stage IV) melanoma;
5. Available blocks for histological examination and/or the subject's consent to undergo biopsy ;
6. Consent to the evaluation of the PD-L1 status and BRAF V600 mutation status at a central laboratory;
7. ECOG score 0-1;
8. Life expectancy of at least 12 weeks ;
9. Measurable target tumor lesions (at least 1 lesion) according to RECIST 1.1 criteria , confirmed by central independent reviewer;
10. In subjects of childbearing potential, willingness to use reliable contraceptive measures throughout the study, from the signing of the informed consent form and for additional 24 weeks after the administration of the last dose of the investigational product.

Exclusion Criteria:

1. Indications for radical (surgical, radiation) therapy;
2. A history of previous systemic antitumor therapy for unresectable or metastatic melanoma ;
3. Prior therapy with checkpoint inhibitors (e.g., anti-CTLA-4 and/or anti-PD-1/PD-L1/PD-L2 products);
4. Prior therapy with BRAF and MEK protein kinase inhibitors;
5. Use of immunostimulants, monoclonal antibodies and/or colony-stimulating factors within less than 4 weeks prior to randomization in the study;
6. Ocular melanoma;
7. Mucosal melanoma;
8. CNS metastases;
9. Impossibility to determine PD-L1 status and/or BRAF status;
10. Subjects with severe comorbidities, life-threatening acute complications of the primary disease (including massive pleural, pericardial, or peritoneal effusions requiring intervention , pulmonary lymphangitis, bleeding, or organ perforation) at the time of signing the informed consent form;
11. Ongoing concomitant diseases at the time of screening, which increase the risk of severe adverse events during the administration of the study therapy:

    * stable angina, functional class III-IV;
    * unstable angina or a history of myocardial infarction within less than 6 months prior to signing the informed consent form;
    * moderate to severe heart failure (classes III and IV according to NYHA classification);
    * uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg) ;
    * a history of atopic asthma , angioedema;
    * respiratory failure (moderate to severe), grade 3 or 4 chronic obstructive pulmonary disease;
    * any other concomitant diseases (including, but not limited to, metabolic, hematological, renal, hepatic, pulmonary, neurological, endocrine, cardiac, infectious, gastrointestinal disorders), which expose the subject to an unacceptable risk during the study therapy;
12. Known or suspected systemic autoimmune diseases (including, but not limited to, systemic lupus erythematosus, Crohn's disease, nonspecific ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, etc.) ;
13. History of interstitial pulmonary disease or pneumonitis requiring systemic glucocorticoids;
14. The need for glucocorticoid therapy (at >10 mg/day prednisolone equivalent doses) or any other drugs with immunosuppressive effects within 14 days prior to randomization;
15. Hematologic abnormalities :

    * neutrophils <1.5×109/L;
    * platelets <100×109/L;
    * hemoglobin <90 g/L;
16. Renal impairment: creatinine ≥2.5×ULN;
17. Hepatic impairment :

    * total bilirubin ≥3×ULN (except for subjects with Gilbert's syndrome, in whom bilirubin levels should not exceed 50 μmol/L),
    * AP, AST or ALT ≥2.5×ULN (≥5×ULN in case of subjects with liver metastases);
18. Any antitumor treatment within less than 4 weeks or surgery within less than 28 days prior to randomization within the study;
19. History of oncological disease, except for radically treated diseases with remission for over 5 years prior randomization in this study ;
20. Conditions limiting the subject's ability to comply with the Protocol requirements (in the Investigator's opinion );
21. Participation in other clinical studies within less than 30 days prior to randomization and during this clinical study ;
22. Acute infections or activation of chronic infectious diseases or systemic antibacterial therapy within less than 28 days prior to randomization;
23. Active hepatitis B, active hepatitis C (confirmed by PCR), active syphilis, HIV-infection, currently or previously ;
24. Impossibility to administer the investigational product intravenously;
25. Impossibility to administer intravenous contrast agents (including due to hypersensitivity to contrast media);
26. Hypersensitivity to any of the components of BCD-100 or BCD-217;
27. A history of hypersensitivity to monoclonal antibody products;
28. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months

SECONDARY OUTCOMES:
Overall survival | 24 months
Overall response rate (partial response + complete response rate) | 24 months
Disease control rate (stable disease + partial response + complete response rate) | 24 months
Time to response | 24 months
Duration of response | 24 months
The proportion of subjects experiencing adverse events related to study therapy | 24 months
The proportion of subjects experiencing any grade 3 or higher adverse events | 24 months
The proportion of subjects with SAEs | 24 months
The proportion of subjects with immune-related adverse events of any severity | 24 months
The proportion of subjects with severe immune-related adverse events | 24 months
The proportion of subjects requiring treatment discontinuation due to AEs | 24 months
The proportion of BAb and NAb positive subjects | 24 months
Ctrough (plasma concentration of anti-PD-1/CTLA-4 monoclonal antibody measured at the end of the dosing interval before the next dose) | 24 months

CONTACTS AND LOCATIONS:
Locations (63):
- Belarus (8):
  - Healthcare Institution "Bobruisk Interdistrict Oncological Dispensary", Babruysk
  - Healthcare Institution "Brest Regional Oncological Dispensary", Brest
  - Health care institution "Grodno University Clinic", Grodno
  - Health Institution "Gomel Regional Clinical Oncology Center", Homyel
  - State Institution "Republican Scientific and Practical Center of Oncology and Medical Radiology named after A.I. N.N. Alexandrov", Lesnoy
  - Healthcare Institution "Minsk City Clinical Cancer Center", Minsk
  - State Institution "Mogilev Regional Oncological Dispensary", Mogilev
  - Healthcare Institution "Vitebsk Regional Clinical Oncology Center", Vitebsk
- India (12):
  - Fortis Hospital, Faridabad
  - Kasturba Medical College and Hospital, Mangalore
  - TATA Memorial Hospital, Mumbai
  - HealthCare Global Enterprises Ltd, NCHRI Cancer Center, Nagpur
  - HealthCare Global Enterprises Ltd Manavata cancer Centre, Nashik
  - Sankalp Superspeciality Hospital, Nashik
  - All India Institute of Medical Science, New Delhi
  - Deenanath Mangeshkar Hospital & Research Center, Pune
  - PDEAS Ayurved Rugnalaya & Steriling Multispeciality Hospital, Pune
  - Horizon Mulitispeciality Hospital, Sangli
  - Shalby Hospital, Surat
  - Kiran Multispeciality hospital &Research, Sūrat
- Russia (43):
  - Chelyabinsk Regional Clinical Center for Oncology and Nuclear Medicine, Chelyabinsk, Chelyabinsk Oblast
  - LLC "New Clinic", Pyatigorsk, Stavropol Kray
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - Regional State Budgetary Institution of Health Care "Altai Regional Oncological Dispensary", Barnaul
  - Limited Liability Company "EVIMED", Chelyabinsk
  - Private healthcare institution "Clinical hospital "RZD-Medicine" of the city of Chelyabinsk", Chelyabinsk
  - State budgetary healthcare institution Leningrad Regional Clinical Hospital, Gatchina
  - State Autonomous Health Institution "Republican Clinical Oncology Dispensary of the Ministry of Health of the Republic of Tatarstan named after Professor M.Z. Sigal", Kazan'
  - State budgetary health care institution "Kuzbass clinical oncological dispensary named after M.S. Rappoport", Kemerovo
  - Regional Goverment Budgetary Healthcare State "Kostroma Oncology Center", Kostroma
  - State Budgetary Institution of Healthcare "Leningrad Regional Clinical Oncological Dispensary named after V.I. L.D. Romana", Kuz'molovskiy
  - "Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - Branch of Hadassah Medical LTD Limited Liability Company, Moscow
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Joint Stock Company "K31 City", Moscow
  - JSC "Medsi Group", Moscow
  - Moscow City Oncology Hospital No. 62, Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Oncology Hospital No. 1 of the Department of Health of the City of Moscow", Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "Moscow Multidisciplinary Clinical Center "Kommunarka" of the Department of Health of the City of Moscow", Moscow
  - Nizhny Novgorod Region State Budgetary Healthcare Facility "Clinical Diagnostics Center", Nizhny Novgorod
  - LLC "DobroMed", Novosibirsk
  - State Budgetary Healthcare Institution "Novosibirsk Regional Clinical Oncology Center" of the Novosibirsk Region, Novosibirsk
  - Federal State Budgetary Institution "National Medical Research Center for Radiology" of the Ministry of Health of the Russian Federation, Obninsk
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Center", Omsk
  - Federal State Budgetary Institution "National Medical Research Center of Oncology named after N.N. Petrov" of the Ministry of Health of the Russian Federation (FSBI "N.N. Petrov National Medical Research Center of Oncology" of the Ministry of Health of Ru, Pesochnyy
  - LLC "Clinical Trials", Saint Petersburg
  - JSC "Modern Medical Technologies", Saint Petersburg
  - City Hospital #40, Kurortny district, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Saint Petersburg State University", Saint Petersburg
  - Federal State Budgetary Health Institution St. Petersburg Clinical Hospital of the Russian Academy of Sciences, Saint Petersburg
  - Limited Liability Company "EuroCityClinic", Saint Petersburg
  - Limited Liability Company "Oncological Research Center", Saint Petersburg
  - Limited Liability Company "Stepmed Clinic", Saint Petersburg
  - Limited Liability Company "Strategic Medical Systems", Saint Petersburg
  - LLC "AV medical group", Saint Petersburg
  - N.N. Petrov National Medicine Research Center of oncology, Saint Petersburg
  - Private Medical Institution Evromedservis, Saint Petersburg
  - State budgetary health care institution "St. Petersburg Clinical Scientific and Practical Center of Specialized Medical Assistance (Oncological)", Saint Petersburg
  - Private institution educational organization of higher education "Medical University "Reaviz", Samara
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - Oncology Dispensary 2, Sochi
  - State Health Care Institution "Volgograd Regional Clinical Oncology Dispensary № 1", Volgograd
  - State Regional Budgetary Healthcare Institution "Regional Clinical Oncology Hospital" of the Yaroslavl Region, Yaroslavl